CLINICAL TRIAL: NCT00972023
Title: A Pilot Study of Androgen Receptor as a Target for the Treatment of ER-/PR-/AR + Breast Cancer
Brief Title: DHEA in Treating Women Undergoing Surgery for Stage I, Stage II, or Stage III Breast Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000653162; P30CA022453 (NIH); WSU-2008-012
Record Dates: First submitted 2009-09-03; First posted 2009-09-04 (Estimated); Results first posted 2013-07-10 (Estimated); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Breast Cancer
Keywords: triple-negative breast cancer; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Dehydroepiandrosterone

ARMS (1):
- DHEA, surgical resection (Experimental): Day-14 (approx. 2 wks prior to surgery): begin a 2 week course of DHEA; Day-7 (approx. 1 wk after starting treatment): answer question about pill diary; Day 0 (approx. 2 wks after starting treatment, within 48 hours prior to surgery;
  Interventions: Drug: DHEA; Procedure: Surgical resection

INTERVENTIONS:
Drug: DHEA — DHEA administration will begin approxiately 14 days prior to surgery.
  Other Names: therapeutic dehydroepiandrosterone
Procedure: Surgical resection — Surgical procedure of the invasive breast cancer

SUMMARY:
RATIONALE: Dehydroepiandrosterone (DHEA) may slow the growth of tumor cells and be an effective treatment for women with breast cancer.

PURPOSE: This phase I trial is studying how well DHEA works in treating women undergoing surgery for stage I, stage II, or stage III breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To identify the effect of the adrenal steroid, dehydroepiandrosterone (DHEA), on tumor proliferation in women with estrogen receptor-negative, progesterone receptor-negative, HER2/neu-negative, and androgen receptor (AR)-positive stage I-III adenocarcinoma of the breast.

Secondary

* To study the effect of DHEA on expression of AR in these patients.
* To assess the effect of DHEA on changes in serum estrogen and androgen hormone levels (e.g., estrone, estradiol, testosterone, dihydrotestosterone, DHEA, and DHEA-sulfate) in these patients.
* To assess the toxicity of DHEA in these patients.
* To follow the clinical course of these patients.

OUTLINE: Patients receive oral dehydroepiandrosterone (DHEA) twice daily on days -14 to 0. Patients then undergo surgery on day 1.

Tissue samples are collected at baseline and at the time of surgery for biomarker analysis (androgen receptor, estrogen receptor, progesterone receptor, HER2/neu, Ki-67, and p53) by IHC. Blood samples are collected at baseline and after completion of treatment with DHEA for analysis of serum hormone (e.g., estrone, estradiol, testosterone, dihydrotestosterone, DHEA, and DHEA-sulfate) and cytokine levels.

After completion of study therapy, patients are followed up at 1 week and then every 6 months for 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed invasive adenocarcinoma of the breast

  * Stage I (T1c), II, or III disease (AJCC staging system)

    * Lesion ≥ 1 cm on breast imaging studies (mammogram, ultrasound, or MRI)
* HER2/neu-negative tumor
* Planning to receive dehydroepiandrosterone (DHEA) prior to surgery
* Disease amenable to surgery with curative intent

  * Scheduled to undergo surgery immediately after completion of DHEA
* No locally advanced or metastatic disease not amenable to surgery
* Hormone receptor status:

  * Estrogen receptor- and progesterone receptor-negative tumor
  * Androgen receptor-positive tumor

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* ECOG performance status (PS) 0-2 OR Karnofsky PS 60-100%
* ANC ≥ 1,000/mm^3
* Platelet count ≥ 75,000/mm^3
* AST and ALT ≤ 2.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2.5 times ULN
* Bilirubin ≤ 2 times ULN
* Hemoglobin > 9 g/dL
* Creatinine normal OR creatinine clearance ≥ 60 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 1 week after completion of study therapy
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to DHEA or anastrozole
* No concurrent uncontrolled illness, including but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness or social situation that would limit compliance with study requirements

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 5 years since prior surgery, radiotherapy, biological therapy, hormone therapy, and/or chemotherapy for invasive breast cancer
* No other concurrent antineoplastic or antitumor agents
* No other concurrent investigational agents

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2010-02; Primary Completion 2010-03 (Actual); Study Completion 2010-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zeina Nahleh, MD, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States

REFERENCES:
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — http://cancer.gov/clinicaltrials

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Cancer center clinic
Groups:
- DHEA, Surgical Resection: DHEA, surgical resection:
  Day-14 (approx. 2 wks prior to surgery): begin a 2 week course of DHEA; Day-7 (approx. 1 wk after starting treatment): answer question about pill diary; Day 0 (approx. 2 wks after starting treatment, within 48 hours prior to surgery;
  DHEA: Administration will begin approxiately 14 days prior to surgery.
  Surgical resection: Surgical procedure of the invasive breast cancer
Period: Overall Study
Arm/Group | DHEA, Surgical Resection
Started | 1
Completed | 0
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- DHEA, Surgical Resection: Day-14 (approx. 2 wks prior to surgery): begin a 2 week course of DHEA; Day-7 (approx. 1 wk after starting treatment): answer question about pill diary; Day 0 (approx. 2 wks after starting treatment, within 48 hours prior to surgery;
  DHEA : DHEA administration will begin approxiately 14 days prior to surgery.
  Surgical resection : Surgical procedure of the invasive breast cancer
Arm/Group | DHEA, Surgical Resection
Number analyzed (Participants) | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Tumor Proliferation (Percentage of Ki-67 Positive Cells)
Time Frame: Baseline, prior to DHEA treatment, within 48 hours prior to surgery and after 14 days of DHEA treatment.
Population: Per protocol, although no analysis was completed, patient chose to receive neoadjuvant chemo instead of surgery & refused follow up.
Arm/Group | DHEA, Surgical Resection
Number analyzed (Participants) | 0

2. Secondary Outcome: Effect of Dehydroepiandrosterone (DHEA) on Androgen Receptor Expression
Time Frame: Baseline, prior to DHEA treatment, within 48 hours prior to surgery and after 14 days of DHEA treatment.
Population: as for outcome 1
Arm/Group | DHEA, Surgical Resection
Number analyzed (Participants) | 0

3. Secondary Outcome: Effect of DHEA on Changes in Serum Estrogen and Androgen Hormone Levels (e.g., Estrone, Estradiol, Testosterone, Dihydrotestosterone, DHEA, and DHEA-sulfate)
Time Frame: Baseline, prior to DHEA treatment, within 48 hours prior to surgery and after 14 days of DHEA treatment.
Population: as for outcome 1
Arm/Group | DHEA, Surgical Resection
Number analyzed (Participants) | 0

4. Secondary Outcome: Toxicity
Time Frame: Within 48 hours prior to surgery and after 14 days of DHEA treatment.
Population: as for outcome 1
Arm/Group | DHEA, Surgical Resection
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | DHEA, Surgical Resection
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No